CLINICAL TRIAL: NCT05429801
Title: Efficacy of Ozone Therapy in Patients With Ankylosing Spondylitis: A Randomized Controlled Study
Brief Title: Ozone Therapy in Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hakan Alkan, Clinical Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60116787-020/14061
Record Dates: First submitted 2022-06-13; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Ankylosing Spondylitis
Keywords: ozone therapy; complementary treatment
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone Therapy (Experimental): Rectal ozone treatment along with medical treatment was administered to the patients in this group, in increasing doses for 5 sessions per week, 20 sessions in total for 4 weeks.
  Interventions: Other: Ozone therapy
- Control group (Active Comparator): The patients in this group continued only their current medical treatment.
  Interventions: Other: Ozone therapy

INTERVENTIONS:
Other: Ozone therapy — Rectal ozone treatment along with standard medical treatment was administered to the patients, in increasing doses for 5 sessions per week, 20 sessions in total for 4 weeks. First week: 25 mg/l, 100 ml; second week: 30 mg/l, 150 ml; third week: 35 mg/l, 200 ml; fourth week: 40 mg/l, 200 ml rectal ozone treatment was applied.

SUMMARY:
The aim of this study was to investigate the effects of rectal ozone therapy added to medical treatment on pain severity, disease activity, spinal mobility, functional status, enthesitis, and quality of life (QoL) in patients with ankylosing spondylitis (AS).

Patients and methods: Patients who fulfilled the modified New York criteria for AS were included in this randomized controlled study. Thirty patients selected according to inclusion and exclusion criteria were randomized into two groups. Rectal ozone treatment along with medical treatment was administered to the patients in group 1, in increasing doses for 5 sessions per week, 20 sessions in total for 4 weeks. The patients in group 2 continued only their current medical treatment. All patients received a comprehensive rheumatologic assessment including pain severity, disease-specific instruments for disease activity, functional status, spinal mobility, enthesitis score, and QoL.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as AS according to the Modified New York criteria

Exclusion Criteria:

* having other concomitant rheumatic diseases,
* receiving anti-TNF-α therapy within the last 3 months,
* being in clinical remission with standard medical treatment,
* being pregnant,
* having diseases such as favism, asthma, pancreatitis, and uncontrolled hyperthyroidism for which ozone therapy is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | Change from baseline VAS at the 4th week after the treatment
  The patients were assessed for low back pain level according to the 10 cm visual analogue scale (VAS) from 0 (no pain) to 10 (maximum pain).

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index | Change from baseline Bath Ankylosing Spondylitis Disease Activity Index at the 4th week after the treatment
  Bath Ankylosing Spondylitis Disease Activity Index was used to assess disease acticvity.The Bath Ankylosing Spondylitis Disease Activity Index has a range of 0 to 10; a lesser number represents less severe disease activity
Ankylosing Spondylitis Disease Activity Score | Change from baseline Ankylosing Spondylitis Disease Activity Score at the 4th week after the treatment
  Ankylosing Spondylitis Disease Activity Score is a new composite index to assess disease activity which contains low back pain, global assessment of the patient, peripheral joint pain and swelling, duration of morning stiffness, and acute phase response parameters.Four disease activity states were chosen by consensus: inactive disease, moderate, high, and very high disease activity. The three cut-offs selected to separate these states were: 1.3, 2.1 and 3.5 units. Hihger score means higher disease activity.
Bath Ankylosing Spondylitis Functional Index | Change from baseline Bath Ankylosing Spondylitis Functional Index at the 4th week after the treatment
  The Bath Ankylosing Spondylitis Functional Index (BASFI) was used to determine the degree of functional limitation in patient with AS. The Bath Ankylosing Spondylitis Functional Index has a score between 0 and 10, with a higher score indicating more functional limitation
Ankylosing Spondylitis Quality of Life | Change from baseline Ankylosing Spondylitis Quality of Life score at the 4th week after the treatment
  The disease-specific instrument Ankylosing Spondylitis Quality of Life (ASQoL) includes 18 yes or no questions related to the impact of disease on sleep, mood, motivation, coping, activities of daily living, independence, relationships, and social life with a total score of 0-18. Lower ASQoL scores represent a better QoL

CONTACTS AND LOCATIONS:
Overall Officials: Füsun Ardıç, Prof, Study Director — Pamukkale University
Locations (1):
- Hakan Alkan, Denizli, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No